CLINICAL TRIAL: NCT06739265
Title: A Phase I/II Study of Golidocitinib in Combination with CHOP in Patients with Newly Diagnosed Peripheral T Cell Lymphoma
Brief Title: Golidocitinib Plus CHOP in Newly Diagnosed PTCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-018
Record Dates: First submitted 2024-11-18; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-09

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- G-CHOP arm (Experimental)
  Interventions: Drug: Golidocitinib plus CHOP

INTERVENTIONS:
Drug: Golidocitinib plus CHOP — Phase 1: dose escalation phase. Drug Golidocitinib: 2 dose level of 150 mg qod and 150 mg qd; CHOP regimen: cyclophosphamide (750 mg/m2 intravenously on day 1), epirubicin (70 mg/m2 intravenously on day 1), vindesine (4 mg intravenously on day 1), and prednisone (60 mg/m2 orally on days 1-5) in a 3-week cycle. Phase 2: dose expansion phase. Drug Golidocitinib: RP2D established in the phase I study; CHOP regimen: cyclophosphamide (750 mg/m2 intravenously on day 1), epirubicin (70 mg/m2 intravenously on day 1), vindesine (4 mg intravenously on day 1), and prednisone (60 mg/m2 orally on days 1-5) in a 3-week cycle.

SUMMARY:
This is single-arm phase I/II study designed to evaluate the safety and efficacy of golcadotinib in combination with the CHOP regimen for patients with newly diagnosed peripheral T-cell lymphoma (PTCL). The study adopts a two-stage design, consisting of a Phase I and a Phase II parts. In the phase I study, a standard "3+3" design will be used. The primary endpoints of the Phase I study are the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D). The primary endpoint of the Phase II study is the complete response rate (CRR) of the golcadotinib combined with CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years;
* Histopathologically confirmed diagnosis of PTCL of one of the following subtypes: (1) Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS); (2) Angioimmunoblastic T-cell lymphoma (AITL); (3) Anaplastic large cell lymphoma (ALCL); or (4) other PTCL subtypes considered eligible by the investigator;
* Patients must have at least one measurable lesion according to the Lugano 2014 criteria: For lymph node lesions, the measurable lymph node must have a long diameter >1.5 cm; for non-lymph node lesions, the measurable extranodal lesion must have a long diameter >1.0 cm;
* ECOG performance status score of 0-3;
* Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count (PLT) ≥75×10^9/L, and hemoglobin (HGB) ≥90 g/L (for patients with bone marrow involvement, ANC can be relaxed to ≥1.0×10^9/L, PLT to ≥50×10^9/L, and HGB to ≥75 g/L);
* Adequate organ function: alanine aminotransferase (ALT) <3 times the upper limit of normal (ULN), total serum bilirubin (TBIL) ≤1.5 times ULN, creatinine clearance ≥50 mL/min, and left ventricular ejection fraction (LVEF) ≥50% as determined by echocardiography.

Exclusion Criteria:

* Extranodal NK/T-cell lymphoma;
* History of acute myocardial infarction or unstable angina, congestive heart failure, symptomatic arrhythmias, or significant QT interval prolongation (men >450 ms, women >470 ms) within the past 6 months;
* Uncontrolled active infection;
* ANC ≤0.5×10^9/L, lymphocyte count ≤0.4×10^9/L, PLT ≤75×10^9/L, ALT ≥3 times the ULN, or creatinine clearance ≤50 mL/min;
* Presence of primary or secondary central nervous system (CNS) lymphoma at the time of enrollment;
* Pregnant or breastfeeding women;
* Patients who have received any investigational drug or radiotherapy within the past 4 weeks;
* Individuals deemed unsuitable for participation by the investigator;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of phase 1 study | 4 weeks since the date of first dose]
  Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) will be established according to the incidence of dose-limiting toxicities (DLTs) of escalated doses of golidocitinib
complete remission rate (CRR) of the phase 2 study | Responses were evaluated after 3 cycles of induction and 1 month after the completion of study therapy (each cycle is 21 days)
  Treatment responses were assessed according to the 2014 Lugano classification criteria.

SECONDARY OUTCOMES:
Progression-free survival | From date of enrollment until documented disease progression or death of any reason (up to 3 years)
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, or death from any cause, whichever occurred first.
Overall survival | From date of enrollment until documented death of any reason (up to 3 years)
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
adverse events | From enrollment till 28 days post the last induction cycle
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Objective Response Rate (ORR) | Responses were evaluated after 3 cycles of induction and 1 month after the completion of study therapy (each cycle is 21 days)
  The ORR was defined as the proportion of patients with CR or PR.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided